CLINICAL TRIAL: NCT03980652
Title: Cheetah - a Cluster Randomized Trial of Sterile Glove and Clean Instrument Change at the Time of Wound Closure to Reduce Surgical Site Infection (SSI). A Trial in Low and Middle Income Countries (LMICs) and A Trial in High Income Countries (HICs)
Brief Title: Cheetah - Sterile Glove and Clean Instrument Change at the Time of Wound Closure to Reduce Surgical Site Infection
Acronym: Cheetah
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1234
Record Dates: First submitted 2019-06-03; First posted 2019-06-10 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: Cluster randomised controlled trial
Who Masked: Participant
Masking Description: The Randomisation is at the hospital level and hospitals will be randomised to the intervention (of separating sterile surgical instruments and gloves at the time of wound closure). Patients will not be made aware of the hospital/theatre randomisation, as patients would also not be aware of the specifics of any operation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Other): Change of gloves and use of separate, sterile instruments before closing the abdominal wall
  Interventions: Procedure: Change of gloves and sterile instruments
- Current routine hospital practice (No Intervention): No change of gloves or use of separate, sterile instruments before closing the abdominal wall

INTERVENTIONS:
Procedure: Change of gloves and sterile instruments — Change of gloves and use of separate , sterile instruments before closing the abdominal wall
  Arms: Intervention

SUMMARY:
To assess whether the practice of using separate sterile gloves and instruments to close wounds at the end of surgery compared to current routine hospital practice can reduce surgical site infection

DETAILED DESCRIPTION:
Internal Pilot

The aim of the 12-month internal pilot is to assess:

1. whether hospitals adhere to their allocation
2. what proportion of patients who are eligible for ChEETAh can be followed up successfully at 30 days after their surgery

Main Study

To assess whether the practice of using separate sterile gloves and instruments to close wounds at the end of surgery compared to current routine hospital practice can reduce surgical site infection at 30-days post-surgery for patients undergoing clean-contaminated, contaminated or dirty abdominal surgery

ELIGIBILITY:
Inclusion Criteria

* Countries: LMICs defined by the Development Assistance Committee (DAC) Official Development Assistance (ODA) list where there are at least 4 eligible hospitals per country in HIC-CHEETAH protocol (HICs are those that do not appear on the Organisation for Economic Co-operation and Development's Official Development Assistance (ODA) list
* Hospitals (clusters): in LMICs where glove and instrument change is not currently routine hospital practice
* Participants: Patients undergoing abdominal surgery who satisfy the following criteria are eligible:
* Emergency (surgery on an unplanned admission) or elective (surgery on a planned admission)
* Intraoperative finding of clean-contaminated, contaminated or dirty surgery
* with at least one abdominal incision that is ≥5cm
* Aged 16 years and over on the day of surgery (applicable to HIC-CHEETAH protocol only)

Participant Exclusion Criteria:

• Patients undergoing caesarean section

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12800 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Surgical Site Infection (SSI) at 30-days post-surgery | 30-days post-surgery
  The Centre for Disease Control (CDC) definition will be used in ChEETAh to identify deep incisional or superficial incisional SSIs

SECONDARY OUTCOMES:
SSI before discharge from hospital | up to 30 days
  SSI will be assessed following the index operation, at the point of discharge, and assessed according to the Centre for Disease Control (CDC) criteria
Re-admission | within 30-days post-surgery
  Unexpected re-admission into hospital for a wound-related problem within 30-days post surgery
Length of hospital stay | Length of hospital stay for the index operation and assessed at the point of discharge up to 30 days
  Length of hospital stay following surgery
Return to normal activities e.g (work, school, or family duties) | The assessment will be made up to 30-days from the index operation.
  Return to normal activities from the date of the index operation will be assessed by a questionnaire via telephone and analysed by the Centre for Disease Control (CDC) criteria.
Death | within 30 days post-surgery
  within 30 days of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mr Aneel Bhangu, Principal Investigator — University of Birmingham

REFERENCES:
- [Derived] NIHR Global Health Research Unit on Global Surgery. Study protocol for a cluster randomised trial of sterile glove and instrument change at the time of wound closure to reduce surgical site infection in low- and middle-income countries (CHEETAH). Trials. 2022 Mar 9;23(1):204. doi: 10.1186/s13063-022-06102-5. PMID 35264227